CLINICAL TRIAL: NCT07160322
Title: Prognosis and Clinical Outcomes of Refractory Dyspnea in Chronic Obstructive Pulmonary Disease: Prospective Observational Study
Brief Title: Refractory Breathlessness in COPD
Acronym: RB-COPD
Status: Recruiting | Type: Observational
Sponsor: Seoul National University (Other)
Responsible Party: Principal Investigator, Hyun Woo Lee, Assistant professor, Seoul National University
Other Study IDs: 2024-0434
Record Dates: First submitted 2025-07-20; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-07

CONDITIONS: COPD
Keywords: Chronic Obstructive Pulmonary Disease (COPD); Refractory Breathlessness; Persistent Dyspnea; Treatment Resistance; Unresponsive to Therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD patients with refractory breathlessness despite LABA/LAMA therapy: Patients with COPD who continue to experience clinically significant dyspnea (mMRC ≥ 2 or CAT ≥ 10) despite at least 3 months of treatment with dual long-acting bronchodilator therapy (LABA/LAMA), showing less than a 1-point reduction in mMRC or less than a 4-point reduction in CAT scores compared with baseline.

SUMMARY:
This study aims to investigate the prognosis and clinical outcomes of patients with chronic obstructive pulmonary disease (COPD) who continue to experience refractory dyspnea despite treatment with long-acting beta-agonist (LABA) and long-acting muscarinic antagonist (LAMA). The research will prospectively follow a cohort of patients to identify clinical factors, lung function parameters, imaging features, and cardiovascular indicators associated with poor treatment response. By comparing these patients with those who show symptom improvement, the study seeks to determine predictors of exacerbations, lung function decline, and mortality. Findings are expected to guide the development of targeted strategies to improve the management of refractory dyspnea in COPD.

DETAILED DESCRIPTION:
The study aims to identify actionable clinical factors and develop predictive models that can enhance personalized management approaches for patients with refractory dyspnea in COPD.

This is a prospective observational cohort study designed to characterize patients with COPD who remain symptomatic despite standard inhaled therapy with LABA/LAMA combination. Participants will be enrolled from outpatient clinics and followed over time to assess changes in respiratory symptoms, lung function, exercise capacity, acute exacerbation frequency, and survival.

Key assessments include:

* Baseline demographic and clinical data (e.g., respiratory symptoms, comorbidities, smoking history).
* Pulmonary function tests (spirometry and lung volumes), exercise capacity evaluations, echocardiography, chest radiographs, and computed tomography (CT).
* Biomarker analysis (blood tests including inflammatory and cardiac markers).

Patients will be classified into two groups:

* Refractory COPD group - Patients with minimal improvement in dyspnea (defined as modified Medical Research Council (mMRC) ≥ 2 with <1 point reduction or COPD Assessment Test (CAT) ≥ 10 with <4 point reduction after ≥3 months of LABA/LAMA therapy).
* Control group - Patients showing symptomatic improvement with the same therapy (mMRC <2 or ≥1 point reduction, or CAT <10 or ≥4 point reduction).

The primary analyses will explore clinical and physiological predictors of poor outcomes, using advanced statistical modeling such as linear mixed-effects models for longitudinal lung function trends, negative binomial regression for exacerbation risk, and Cox proportional hazards models for survival analysis.

Assessments:

Baseline and follow-up evaluations will include demographic and clinical data, comorbidities, smoking history, inhaler adherence and technique, spirometry, lung volume measurements, 6-minute walk tests, echocardiography, chest radiographs, and high-resolution CT scans. Blood tests will include complete blood count, inflammatory markers (C-reactive protein (CRP), fibrinogen), N-terminal pro-B-type natriuretic peptide (NT-proBNP), and cardiac enzymes.

Statistical Analysis:

Longitudinal trends: Changes in lung function, symptoms, and exercise capacity will be assessed using linear mixed-effects models to evaluate the influence of clinical factors.

Acute exacerbations: The frequency of moderate-to-severe exacerbations will be analyzed using negative binomial regression or zero-inflated models when appropriate.

Mortality: Logistic regression will estimate 1-, 3-, and 5-year mortality risk, while Cox proportional hazards models will evaluate time-to-event outcomes.

Predictive modeling: Candidate biomarkers and imaging features will be incorporated into multivariable predictive models to identify key determinants of poor prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years) diagnosed with chronic obstructive pulmonary disease (COPD) according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2025 criteria:
* Presence of COPD risk factors (e.g., smoking history, occupational exposure, genetic predisposition).
* Typical symptoms such as dyspnea, cough, or sputum production.
* Post-bronchodilator FEV1/FVC < 0.70.
* Regular outpatient follow-up at the respiratory clinic.
* Received LABA/LAMA combination therapy for at least 3 months prior to enrollment.
* Ability and willingness to provide written informed consent.

Exclusion Criteria:

* Poor adherence to LABA/LAMA therapy (medication possession rate < 50%) or refusal of treatment.
* Inability or unwillingness to comply with scheduled visits, examinations, or follow-up procedures.
* Presence of severe comorbid conditions expected to significantly affect prognosis, including:

  * End-stage diseases with life expectancy < 1 year.
  * Terminal malignancies receiving hospice or palliative care.
* Any condition that, in the opinion of the investigator, would interfere with study participation or data reliability.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll adult patients (≥ 18 years) diagnosed with chronic obstructive pulmonary disease (COPD) according to the GOLD 2025 criteria, who are receiving combination therapy with long-acting beta2-agonist (LABA) and long-acting muscarinic antagonist (LAMA). Participants include both patients who continue to experience refractory dyspnea despite treatment and those who show symptomatic improvement. All participants must be able to attend regular outpatient visits and provide written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 730 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Annual rate of acute exacerbations in COPD | Up to 5 years (annualized rate)
  Annualized rate of moderate-to-severe exacerbations per patient-year, defined as episodes requiring systemic corticosteroids, antibiotics, or hospitalization.
  Moderate exacerbations will be defined as events requiring treatment with systemic corticosteroids and/or antibiotics without hospitalization. Severe exacerbations will be defined as events leading to hospitalization or emergency department visit.
  Unit: Number of exacerbations per patient-year
All-cause mortality | 1-, 3-, and 5-year follow-up.
  Proportion of participants who die from any cause Unit: Percentage of participants (%) or Number of deaths

SECONDARY OUTCOMES:
Annual forced expiratory volume in one second (FEV1) decline rate | Baseline and annually for up to 5 years.
  Rate of change in forced expiratory volume in one second (FEV1) (Milliliters per year (mL/year)) measured by spirometry Annual decline in FEV1 will be assessed using linear mixed-effects models.
Annual forced expiratory volume in one second to forced vital capacity ratio (FEV1/FVC ratio) decline rate | Baseline and annually for up to 5 years.
  Rate of change in post-bronchodilator forced expiratory volume in one second to forced vital capacity (FEV1/FVC ) ratio (%/year) measured by spirometry Annual decline in FEV1/FVC will be assessed using linear mixed-effects models.

OTHER OUTCOMES:
Change in modified Medical Research Council (mMRC) dyspnea scores from baseline | Baseline, 3-6 months, and annually for up to 5 years.
  Mean change in mMRC score from baseline Unit: Score units (0-4 scale)
Change in CAT scores from baseline | Baseline, 3-6 months, and annually for up to 5 years.
  Mean change in CAT score from baseline Unit: Score units (0-40 scale)
Change in Charlson Comorbidity Index (CCI) from baseline | Baseline and annually for up to 5 years.
  Mean change in CCI score Unit: Score units
Change in COPD-specific Comorbidity Test (COTE) index from baseline | Baseline and annually for up to 5 years.
  Mean change in COTE index Unit: Score units
Change in COPD Comorbidity (COMCOLD) index from baseline | Baseline and annually for up to 5 years.
  Mean change in COMCOLD index Unit: Score units
Change in medication possession rate (MPR) from baseline | Baseline and annually for up to 5 years.
  Mean change in MPR, expressed as % of days with medication available Unit: Percentage (%)
Change in proportion of days covered (PDC) from baseline | Baseline and annually for up to 5 years.
  Mean change in PDC, expressed as % of days with medication available Unit: Percentage (%)
Change in white blood cell (WBC) from baseline | Baseline and annually for up to 5 years.
  Mean change in WBC count from baseline Unit: ×10⁹ cells/L
Change in blood eosinophil count (BEC) from baseline | Baseline and annually for up to 5 years.
  Mean change in BEC from baseline Unit: cells/L
Change in immunoglobulin E (IgE) from baseline | Baseline and annually for up to 5 years.
  Mean change in IgE from baseline Unit: International Units per milliliter (IU/mL)
Change in fibrinogen from baseline | Baseline and annually for up to 5 years.
  Mean change in fibrinogen from baseline Unit: milligrams per deciliter (mg/dL)
Change in cortisol from baseline | Baseline and annually for up to 5 years.
  Mean change in cortisol measured at 8 AM from baseline Unit: micrograms per deciliter (µg/dL)
Change in C-reactive protein (CRP) from baseline | Baseline and annually for up to 5 years.
  Mean change in CRP from baseline Unit: milligrams per liter (mg/L)
Change in N-terminal pro-B-type natriuretic peptide (NT-proBNP) from baseline | Baseline and annually for up to 5 years.
  Mean change in NT-proBNP from baseline Unit: picograms per milliliter (pg/mL)
Change in Troponin I from baseline | Baseline and annually for up to 5 years.
  Mean change in Troponin I from baseline Unit: nanograms per milliliter (ng/mL)
Change in difference between respiratory resistance at 5 Hz and 20 Hz (R5-R20) from baseline | Baseline and annually for up to 5 years.
  Mean change in R5-R20 from baseline Unit: cmH₂O/L/s
Change in resonant frequency (Fres) from baseline | Baseline and annually for up to 5 years.
  Mean change in Fres from baseline Unit: Hertz (Hz)
Change in reactance at 5 Hz (X5) from baseline | Baseline and annually for up to 5 years.
  Mean change in X5 from baseline Unit: cmH₂O/L/s
Change in area of reactance (AX) from baseline | Baseline and annually for up to 5 years.
  Mean change in AX from baseline Unit: cmH₂O/L
Change in parametric response mapping of functional small airway disease (PRMfSAD) in chest CT from baseline | Baseline and annually for up to 5 years.
  Mean change in PRMfSAD from baseline Unit: Percentage of lung volume (%)
Change in low attenuation area in inspiratory chest CT from baseline | Baseline and annually for up to 5 years.
  Mean change in low attenuation area (<-950 Hounsfield unit (HU)) in inspiratory chest CT from baseline Unit: Percentage of lung volume (%)
Change in low attenuation area in expiratory chest CT from baseline | Baseline and annually for up to 5 years.
  Mean change in low attenuation area (<-856 hounsfield unit (HU)) in expiratory chest CT from baseline Unit: Percentage of lung volume (%)
Change in square root of wall area for a theoretical airway with 10 mm internal perimeter (Pi10) in chest CT from baseline | Baseline and annually for up to 5 years.
  Mean change in square root of wall area for a theoretical airway with 10 mm internal perimeter (Pi10) from baseline Unit: millimeters (mm)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University College of Medicine, Seoul Metropolitan Government-Seoul National University Boramae Medical Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the dataset contains sensitive personal health information, and there are no current plans or infrastructure for secure data sharing. Data will be used solely for analyses specified in the approved protocol and will remain confidential in accordance with institutional and IRB guidelines.